CLINICAL TRIAL: NCT04667117
Title: An Open-label Multicenter Study to Assess Response to Influenza Vaccine in Participants With Multiple Sclerosis Treated With Ofatumumab 20 mg Subcutaneously
Brief Title: A Multicenter Study to Assess Response to Influenza Vaccine in Multiple Sclerosis Participants Treated With Ofatumumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GUS12
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: ofatumumab; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Influenza Vaccines; ofatumumab

STUDY DESIGN:
Intervention Model Description: Parallel, prospective study
Masking Description: Unblinded treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients with relapsing multiple sclerosis (MS) receiving a 2020-2021, 2021-2022, or 2022-2023 inactivated influenza vaccine two weeks prior to ofatumumab start
  Interventions: Biological: Quadrivalent influenza vaccine; Drug: Ofatumumab
- Cohort 2 (Experimental): Patients with relapsing MS receiving a 2020-2021, 2021-2022, 2022-2023 inactivated influenza vaccine at least 4 weeks after ofatumumab start
  Interventions: Biological: Quadrivalent influenza vaccine; Drug: Ofatumumab
- Cohort 3 (Active Comparator): Patients with relapsing MS currently on iDMT receiving a 2020-2021, 2021-2022, or 2022-2023 inactivated influenza vaccine
  Interventions: Biological: Quadrivalent influenza vaccine; Drug: iDMT

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — 2020-2021, 2021-2022, or 2022-2023 inactivated quadrivalent influenza vaccine. Participants received the vaccine within 9 calendar days after the Screening Visit, before the Week 0 Visit occurred.
Drug: Ofatumumab — Auto-injector containing 20 mg ofatumumab (20 mg/0.4mL) for subcutaneous (s.c.) administration.
  * Participants in Cohort 1 received loading doses of 20 mg ofatumumab s.c. at Weeks 2, 3, and 4 in the Investigational Period. In the open-label Extension Period, they administered the first dose of ofatumumab at Week 6 and continued monthly dosing until the final dose at Week 26. Novartis supplied participants in Cohort 1 with ofatumumab treatment.
  * Participants in Cohort 2 continued on their commercially prescribed ofatumumab treatment during the Investigational Period. In the open-label Extension Period, they continued to administer ofatumumab monthly until the final dose at Week 28. Cohort 2 participants in the extension could have either remained on their prescribed ofatumumab or switched to study supplied ofatumumab.
  Arms: Cohort 1; Cohort 2
Drug: iDMT — Participants in Cohort 3 continued on their commercially prescribed injectable disease modifying therapy (iDMT) during the Investigational Period.
  Arms: Cohort 3

SUMMARY:
To assess whether participants treated with ofatumumab 20 mg subcutaneous (s.c.) administered once every 4 weeks (q4) can mount an adequate immune response to inactivated influenza vaccine as measured by humoral responses compared to participants on an iDMT.

DETAILED DESCRIPTION:
Vaccinations against influenza are an important part of effective management of multiple sclerosis (MS).

Ofatumumab is a human anti-CD20 monoclonal antibody (mAb) which depletes B-cells, a component of the immune system. This study investigates if ofatumumab treated patients can have an immune response that may be protective after receiving the influenza vaccine.

There were 3 study periods:

* Screening Period of up to 1 week to assess eligibility requirements.
* Investigational Period of 4 weeks All participants received an inactivated influenza vaccine within 9 calendar days after the Screening Visit, before the Week 0 Visit occurred.

Participants in Cohort 1 received loading doses of 20 mg ofatumumab administered subcutaneously (s.c.) at Weeks 2, 3, and 4.

Participants in Cohort 2 continued taking their prescribed ofatumumab as per their dosing schedule throughout the Investigational Period.

Participants in Cohort 3 continued administration of their prescribed injectable disease modifying therapy (iDMT) as per their dosing schedule in the Investigational Period.

• Optional, 6-month open-label Extension Period Participants in Cohort 1 were administered their first dose of ofatumumab at Week 6; thereinafter, they continued monthly dosing until the final dose at Week 26.

Participants in Cohort 2 continued to receive ofatumumab monthly until the final dose at Week 28.

Participants in Cohort 3 did not enter the open-label Extension Period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Age 18-55 years old
3. Diagnosis of relapsing MS by 2017 revised McDonald criteria
4. Must be willing to comply with the study schedule
5. Planning to receive a 2020-2021, 2021-2022, or 2022-2023 inactivated influenza vaccine
6. Planning to start treatment with ofatumumab or already on commercially prescribed ofatumumab for at least 2 weeks prior to the screening visit

   Participants in Cohort 3 must fulfill criteria 1-5 above in addition to the following:
7. Participant must currently be receiving iDMT

Exclusion Criteria:

1. Already has received the 2020-2021, 2021-2022, or 2022-2023 season influenza vaccine
2. Known hypersensitivity to any component of the influenza vaccine
3. Any safety finding including low IgG and/or low IgM levels requiring an ofatumumab treatment interruption within the 12 weeks immediately prior to Week 0
4. Any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks prior to or oral antibiotics within two weeks prior to Week 0
5. Known clinical diagnosis of influenza infection during the 2020-2021 influenza season prior to starting the study based on investigator's or subject's personal physician's judgement (laboratory report of confirmed influenza infection is not required)
6. Prior treatment with B-cell targeted therapies (e.g., rituximab or ocrelizumab), lymphocyte-trafficking blockers, alemtuzumab, anti-CD4, cladribine, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, bone marrow transplantation. Treatment with a natalizumab within 6 months of week 0
7. Treatment with an S1P modulator within 60 days prior to Week 0
8. Participants with any known active systemic bacterial, fungal or viral or fungal infections (such as hepatitis, progressive multifocal leukocencephalopathy, COVID-19 or HIV), or known to have acquired immunodeficiency syndrome (AIDS)
9. Participation in another interventional clinical trial within 14 days prior to the screening visit
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
11. Women of child-bearing potential
12. Patients with a history of Guillain-Barre syndrome within 6 weeks of receiving the influenza vaccination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hope Research Institute Center Neurology and Spine, Phoenix, Arizona
  - Infinity Clinical Research LLC, Hollywood, Florida
  - The MS Center for Innovation in Care, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Steingo B, Subei A, Riser E, Gitt J, Stankiewicz J, Piccolo R, Wyse K, Weinstock-Guttman B. Immune response to influenza vaccine in patients with relapsing multiple sclerosis treated with ofatumumab: Results from an open-label, multicenter, phase 4 study. Mult Scler Relat Disord. 2025 May;97:106382. doi: 10.1016/j.msard.2025.106382. Epub 2025 Mar 8. PMID 40107181
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 3 sites in the United States.
Pre-assignment Details: Participants underwent a screening period of up to 1 week. After screening there was a 4-week investigational period and an optional 6-month open-label extension period.
Period: Investigational Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 22 | 22 | 19
Completed | 22 | 21 | 18
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 1 | 0
Period: Extension Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 22 | 11 | 0
Completed | 21 | 11 | 0
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 22 | 22 | 19 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (8.88) | 38.9 (9.03) | 43.3 (7.12) | 41.1 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 14 | 48
  Male | 3 | 7 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 4 | 4 | 9
  White | 21 | 18 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroprotection at Week 4 (Observed Case)
Description: A seroprotection responder was a participant achieving seroprotection as defined by a post-vaccination hemagglutination inhibition (HI) titer ≥ 40 at Week 4. Seroprotection against ten influenza strains was analyzed. The analysis was performed taking into consideration observed data.
Time Frame: Week 4
Population: Participants in the Safety Set with an available value for the outcome measure. Safety Set included all participants who had received inactivated influenza vaccine and at last 1 dose of study drug. For each influenza strain, the number of participants analyzed corresponds to the participants with both pre-vaccination and post-vaccination HI titers for the corresponding strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 22 | 17
percentage of participants
  Influenza A Brisbane: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Brisbane | 100.00 [47.82 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00]
  Influenza A Cambodia: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Cambodia | 100.00 [75.29 to 100.00] | 80.00 [28.36 to 99.49] | 85.71 [42.13 to 99.64]
  Influenza A Kansas: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Kansas | 100.00 [47.82 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00]
  Influenza A Michigan: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Michigan | 100.00 [47.82 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00]
  Influenza A Singapore: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Singapore | 100.00 [47.82 to 100.00] | 100.00 [15.81 to 100.00] | 100.00 [2.50 to 100.00]
  Influenza A Victoria: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Victoria | 100.00 [75.29 to 100.00] | 100.00 [47.82 to 100.00] | 100.00 [59.04 to 100.00]
  Influenza A Wisconsin: number analyzed (Participants) | 13 | 20 | 16
  Influenza A Wisconsin | 61.54 [31.58 to 86.14] | 40.00 [19.12 to 63.95] | 68.75 [41.34 to 88.98]
  Influenza B Colorado: number analyzed (Participants) | 5 | 2 | 1
  Influenza B Colorado | 60.00 [14.66 to 94.73] | 50.00 [1.26 to 98.74] | 100.00 [2.50 to 100.00]
  Influenza B Phuket | 77.78 [52.36 to 93.59] | 68.18 [45.13 to 86.14] | 76.47 [50.10 to 93.19]
  Influenza B Washington: number analyzed (Participants) | 13 | 5 | 7
  Influenza B Washington | 76.92 [46.19 to 94.96] | 20.00 [0.51 to 71.64] | 71.43 [29.04 to 96.33]

2. Primary Outcome: Percentage of Participants Achieving Seroprotection at Week 4 (Non-responder Imputation)
Description: A seroprotection responder was a participant achieving seroprotection as defined by a post-vaccination hemagglutination inhibition (HI) titer ≥ 40 at Week 4. Seroprotection against ten influenza strains was analyzed. Non-responder imputation (NRI) for missing data was applied.
Time Frame: Week 4
Population: Safety Set including all participants who had received inactivated influenza vaccine and at last 1 dose of study drug. For each influenza strain, the number of participants analyzed corresponds to the participants with pre-vaccination HI titers for the corresponding strain.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 22 | 22 | 19
percentage of participants
  Influenza A Brisbane: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Brisbane | 55.56 [21.20 to 86.30] | 66.67 [9.43 to 99.16] | 100.00 [2.50 to 100.00]
  Influenza A Cambodia: number analyzed (Participants) | 15 | 5 | 9
  Influenza A Cambodia | 86.67 [59.54 to 98.34] | 80.00 [28.36 to 99.49] | 66.67 [29.93 to 92.51]
  Influenza A Kansas: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Kansas | 55.56 [21.20 to 86.30] | 66.67 [9.43 to 99.16] | 100.00 [2.50 to 100.00]
  Influenza A Michigan: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Michigan | 55.56 [21.20 to 86.30] | 66.67 [9.43 to 99.16] | 100.00 [2.50 to 100.00]
  Influenza A Singapore: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Singapore | 55.56 [21.20 to 86.30] | 66.67 [9.43 to 99.16] | 100.00 [2.50 to 100.00]
  Influenza A Victoria: number analyzed (Participants) | 15 | 5 | 9
  Influenza A Victoria | 86.67 [59.54 to 98.34] | 100.00 [47.82 to 100.00] | 77.78 [39.99 to 97.19]
  Influenza A Wisconsin: number analyzed (Participants) | 15 | 20 | 18
  Influenza A Wisconsin | 53.33 [26.59 to 78.73] | 40.00 [19.12 to 63.95] | 61.11 [35.75 to 82.70]
  Influenza B Colorado: number analyzed (Participants) | 9 | 3 | 1
  Influenza B Colorado | 33.33 [7.49 to 70.07] | 33.33 [0.84 to 90.57] | 100.00 [2.50 to 100.00]
  Influenza B Phuket | 63.64 [40.66 to 82.80] | 68.18 [45.13 to 86.14] | 68.42 [43.45 to 87.42]
  Influenza B Washington: number analyzed (Participants) | 15 | 5 | 9
  Influenza B Washington | 66.67 [38.38 to 88.18] | 20.00 [0.51 to 71.64] | 55.56 [21.20 to 86.30]

3. Secondary Outcome: Percentage of Participants Achieving Seroconversion at Week 4 (Observed Case)
Description: Seroconversion was defined as: • a ≥ 4-fold increase in HI titers after vaccination (in participants with pre-vaccination HI titers ≥ 10) OR • post-vaccination HI titers ≥ 40 (in participants with pre-vaccination HI titers < 10) Seroconversion against ten influenza strains was analyzed. The analysis was performed taking into consideration observed data.
Time Frame: Baseline (pre-vaccination), Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 22 | 17
percentage of participants
  Influenza A Brisbane: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Brisbane | 80.00 [28.36 to 99.49] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50]
  Influenza A Cambodia: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Cambodia | 84.62 [54.55 to 98.08] | 20.00 [0.51 to 71.64] | 42.86 [9.90 to 81.59]
  Influenza A Kansas: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Kansas | 40.00 [5.27 to 85.34] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50]
  Influenza A Michigan: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Michigan | 60.00 [14.66 to 94.73] | 0.00 [0.00 to 84.19] | 100.00 [2.50 to 100.00]
  Influenza A Singapore: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Singapore | 40.00 [5.27 to 85.34] | 0.00 [0.00 to 84.19] | 0.00 [0.00 to 97.50]
  Influenza A Victoria: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Victoria | 92.31 [63.97 to 99.81] | 20.00 [0.51 to 71.64] | 42.86 [9.90 to 81.59]
  Influenza A Wisconsin: number analyzed (Participants) | 13 | 20 | 16
  Influenza A Wisconsin | 46.15 [19.22 to 74.87] | 10.00 [1.23 to 31.70] | 37.50 [15.20 to 64.57]
  Influenza B Colorado: number analyzed (Participants) | 5 | 2 | 1
  Influenza B Colorado | 60.00 [14.66 to 94.73] | 0.00 [0.00 to 84.19] | 100.00 [2.50 to 100.00]
  Influenza B Phuket | 50.00 [26.02 to 73.98] | 18.18 [5.19 to 40.28] | 41.18 [18.44 to 67.08]
  Influenza B Washington: number analyzed (Participants) | 13 | 5 | 7
  Influenza B Washington | 38.46 [13.86 to 68.42] | 0.00 [0.00 to 52.18] | 42.86 [9.90 to 81.59]

4. Secondary Outcome: Percentage of Participants Achieving Seroconversion at Week 4 (Non-responder Imputation)
Description: Seroconversion was defined as: • a ≥ 4-fold increase in HI titers after vaccination (in participants with pre-vaccination HI titers ≥ 10) OR • post-vaccination HI titers ≥ 40 (in participants with pre-vaccination HI titers < 10) Seroconversion against ten influenza strains was analyzed. Non-responder imputation (NRI) for missing data was applied.
Time Frame: Baseline (pre-vaccination), Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 22 | 22 | 19
percentage of participants
  Influenza A Brisbane: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Brisbane | 44.44 [13.70 to 78.80] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 97.50]
  Influenza A Cambodia: number analyzed (Participants) | 15 | 5 | 9
  Influenza A Cambodia | 73.33 [44.90 to 92.21] | 20.00 [0.51 to 71.64] | 33.33 [7.49 to 70.07]
  Influenza A Kansas: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Kansas | 22.22 [2.81 to 60.01] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 97.50]
  Influenza A Michigan: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Michigan | 33.33 [7.49 to 70.07] | 0.00 [0.00 to 70.76] | 100.00 [2.50 to 100.00]
  Influenza A Singapore: number analyzed (Participants) | 9 | 3 | 1
  Influenza A Singapore | 22.22 [2.81 to 60.01] | 0.00 [0.00 to 70.76] | 0.00 [0.00 to 97.50]
  Influenza A Victoria: number analyzed (Participants) | 15 | 5 | 9
  Influenza A Victoria | 80.00 [51.91 to 95.67] | 20.00 [0.51 to 71.64] | 33.33 [7.49 to 70.07]
  Influenza A Wisconsin: number analyzed (Participants) | 15 | 20 | 18
  Influenza A Wisconsin | 40.00 [16.34 to 67.71] | 10.00 [1.23 to 31.70] | 33.33 [13.34 to 59.01]
  Influenza B Colorado: number analyzed (Participants) | 9 | 3 | 1
  Influenza B Colorado | 33.33 [7.49 to 70.07] | 0.00 [0.00 to 70.76] | 100.00 [2.50 to 100.00]
  Influenza B Phuket | 40.91 [20.71 to 63.65] | 18.18 [5.19 to 40.28] | 36.84 [16.29 to 61.64]
  Influenza B Washington: number analyzed (Participants) | 15 | 5 | 9
  Influenza B Washington | 33.33 [11.82 to 61.62] | 0.00 [0.00 to 52.18] | 33.33 [7.49 to 70.07]

5. Secondary Outcome: Fold Change From Baseline in Hemagglutination Inhibition Titers
Description: Hemagglutination inhibition (HI) antibody titers were measured in serum samples pre-vaccination (baseline) and post-vaccination (Week 4). The geometric mean of the ratio of post-vaccination to pre-vaccination HI titer was calculated to estimate the average fold change in HI titer after vaccination compared to before vaccination.
Time Frame: Baseline (pre-vaccination), Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio to baseline in HI titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 22 | 17
Ratio to baseline in HI titer
  Influenza A Brisbane: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Brisbane | 5.3 [2.3 to 12.3] | 1.4 [0.0 to 115.6] | 2.0
  Influenza A Cambodia: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Cambodia | 9.4 [4.2 to 21.0] | 1.4 [0.4 to 5.5] | 2.9 [1.1 to 7.7]
  Influenza A Kansas: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Kansas | 2.6 [1.0 to 7.0] | 1.0 [NA to NA] — In instances where SD=0 (because all values were the same), the confidence interval for the geometric mean was not calculated as the limits of the confidence interval are exactly the same as the geometric mean. | 2.0
  Influenza A Michigan: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Michigan | 5.5 [1.1 to 26.8] | 0.9 [0.1 to 5.4] | 4.0
  Influenza A Singapore: number analyzed (Participants) | 5 | 2 | 1
  Influenza A Singapore | 4.3 [0.9 to 20.6] | 1.0 [NA to NA] — In instances where SD=0 (because all values were the same), the confidence interval for the geometric mean was not calculated as the limits of the confidence interval are exactly the same as the geometric mean. | 2.0
  Influenza A Victoria: number analyzed (Participants) | 13 | 5 | 7
  Influenza A Victoria | 8.6 [4.3 to 17.3] | 1.3 [0.5 to 3.5] | 3.6 [1.2 to 11.3]
  Influenza A Wisconsin: number analyzed (Participants) | 13 | 20 | 16
  Influenza A Wisconsin | 4.9 [2.0 to 12.0] | 1.7 [1.0 to 3.0] | 2.6 [1.2 to 5.4]
  Influenza B Colorado: number analyzed (Participants) | 5 | 2 | 1
  Influenza B Colorado | 3.0 [1.1 to 8.1] | 1.4 [0.0 to 115.6] | 4.0
  Influenza B Phuket | 3.8 [2.5 to 5.7] | 1.3 [0.9 to 1.9] | 2.2 [1.0 to 4.6]
  Influenza B Washington: number analyzed (Participants) | 13 | 5 | 7
  Influenza B Washington | 3.5 [1.7 to 7.3] | 0.9 [0.6 to 1.3] | 2.8 [1.3 to 6.0]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), AEs Leading to Discontinuation and Serious Adverse Events (SAEs)
Description: Number of participants with adverse events (any AEs regardless of seriousness), AEs leading to study drug discontinuation and serious adverse events (SAEs). On-study AEs are defined as AEs which started or worsened on or after the date of the visit at Week 0.
Time Frame: From Week 0 to Week 26 (Cohort 1), Week 28 (Cohort 2) and Week 4 (Cohort 3)
Population: Safety Set including all participants who had received inactivated influenza vaccine and at last 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 22 | 22 | 19
Participants
  AEs | 16 | 6 | 2
  AEs leading to study drug discontinuation | 0 | 0 | 0
  SAEs | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From Week 0 to Week 26 (Cohort 1), Week 28 (Cohort 2) and Week 4 (Cohort 3)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22 | 0/19
Other Adverse Events (participants affected / at risk) | 16/22 | 6/22 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=22) | Cohort 2 (N=22) | Cohort 3 (N=19)
Multiple sclerosis pseudo relapse (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=22) | Cohort 2 (N=22) | Cohort 3 (N=19)
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Influenza like illness (General disorders) | 2 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Injury associated with device (General disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 4 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04667117/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04667117/SAP_001.pdf